CLINICAL TRIAL: NCT01429051
Title: A Dose Titrated Clinical Trial With a Placebo-controlled, Double-blind, Randomised, Cross-over Phase to Demonstrate the Efficacy of 400 μg Intranasal Fentanyl (INFS) Dose Strength, and to Evaluate 12 Weeks Safety and Nasal Tolerability of All Dose Strengths Between 50 μg and 400 μg, in Cancer Patients With Breakthrough Pain.
Brief Title: A Clinical Trial With Intranasal Fentanyl in Cancer Patients With Breakthrough Pain
Acronym: NOSE-400
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FT-1301-032-SP; 2010-021096-85 (EudraCT Number); U1111-1133-6364 (Registry Identifier: WHO); 2011/776 (Registry Identifier: REK)
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Break Through Pain; Cancer
Keywords: Break through pain; BTP; Cancer; Intranasal Fentanyl Spray; INFS; cancer patients
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal Fentanyl Spray (INFS) (Experimental): All participants were step-wise titrated to an effective dose of 50, 100, 200 or 400 μg INFS in the Titration Phase (I). Participants titrated to 200 or 400 μg INFS in the Titration Phase were randomized to an 8-spray sequence in the Efficacy Phase (II); 6 BTP episodes were treated with 400 μg INFS and 2 BTP episodes with placebo in a random sequence. Participants entered the Tolerability Phase (III) either directly from the Titration Phase (with an effective dose of 50 or 100 μg) or from the Efficacy Phase (400 μg) and continued with this specific dose, unless adjustment was needed, for a total treatment time of 12 weeks.
  Interventions: Drug: Intranasal Fentanyl Spray (INFS); Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Fentanyl Spray (INFS) — Applied as 1 puff (= 1 dose) in one nostril, or applied as two puffs (= 2 doses, 1 in each nostril) with ten minutes apart.
  Other Names: Instanyl®
Drug: Placebo — Matching intranasal placebo spray

SUMMARY:
The aim of this clinical trial was to demonstrate the efficacy of a 400 μg dose strength of intranasal fentanyl spray (INFS, Instanyl®) and to evaluate the safety and to establish long term tolerability of treatment with INFS doses of 50, 100, 200 and 400 μg.

DETAILED DESCRIPTION:
This is a clinical trial with 12 weeks treatment of Intranasal fentanyl (INFS) in cancer patients with breakthrough pain (BTP). It was composed of a dose titrated, placebo-controlled, double-blind, randomised, cross-over efficacy phase, combined with a titration and a tolerability phase assessing the safety and nasal tolerability of INFS. The trial is set up with a screening period and three treatment phases: a titration phase (I), an efficacy phase (II) and a tolerability phase (III). The entire trial period for each completed patient consisted of the one week screening period and 12 weeks treatment with INFS.

ELIGIBILITY:
Inclusion Criteria:

All inclusion criteria were answered 'yes' for a patient to participate in the clinical trial.

* Is the patient a cancer patient with breakthrough Pain (BTP)?
* Has the patient received either oral opioids or transdermal fentanyl for treatment of background pain (BGP) within the last month prior to the screening visit?
* Is the current dose of prescribed opioids (for BGP) equivalent to 60-1000 mg oral morphine/day?
* Has the patient's BGP for the last 7 days prior to the screening visit been generally stable, and on average controlled to a mild level (defined as ≤ 4 on the 11-point Numerical Rating Scale [NRS])?
* Does the patient (at the time of the screening visit) experience his/her current BTP episodes to be of such severe pain intensity, that he/she in general needs additional analgesia (i.e. on top of the background opioid treatment)?
* Has the patient on average for the last 7 days prior to the screening visit had at least three BTP episodes per week, but no more than four BTP episodes per day?
* Is the patient able to use intranasal drugs?
* Is the life expectancy of the patient at least 3 months from the date of the screening visit?

Exclusion Criteria:

1. Has the patient had an illicit substance abuse within the last year prior to screening?
2. Does the patient have severe hepatic impairment? - defined as alanine aminotransferase (ALT or) aspartate aminotransferase (AST) levels > 3x upper limit of normal (ULN)
3. Does the patient have severe renal impairment? - defined as serum creatinine ≥ 3.0 mg/dl (265 micromol/L)
4. Has the patient ever had facial radiotherapy or is the patient scheduled to facial radiotherapy?
5. Has the patient been treated with any monoamine oxidase (MAO) inhibitors within the last 14 days prior to the screening visit?
6. Does the patient have severe impaired respiratory function, which may increase the risk of clinically relevant respiratory depression by BTP fentanyl treatment?
7. Is the patient known to be hypersensitive to fentanyl or to other opioids or any of their excipients?
8. Does the patient have any head injury, primary brain tumor or other pathological conditions, which could significantly increase the risk of increased intracranial pressure or impaired consciousness?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (11):
- Hungary (5):
  - Budapest
  - Debrecen
  - Kazincbarcika
  - Nyíregyháza
  - Pécs
- Norway (2):
  - Drammen
  - Trondheim
- Russia (4):
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Yaroslavl

REFERENCES:
- [Derived] Thronaes M, Popper L, Eeg M, Jaatun E, Kvitberg M, Kaasa S. Efficacy and tolerability of intranasal fentanyl spray in cancer patients with breakthrough pain. Clin Ther. 2015 Mar 1;37(3):585-96. doi: 10.1016/j.clinthera.2014.12.010. Epub 2015 Jan 30. PMID 25641199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in Hungary, Norway and Russia from 08 August 2011 to 04 January 2013.
Pre-assignment Details: The first dose of Intranasal Fentanyl Spray (INFS) was taken at the clinic for training purposes and was not related to treatment of a BTP episode. One patient received the initial 50 μg test dose but did not receive INFS for titration, but is included in the safety analysis set.
Period: Titration Phase
Arm/Group | Intranasal Fentanyl Spray (INFS)
Started | 45
Completed | 33
Not Completed | 12
Not completed — Death | 1
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 1
Not completed — Unsuccessful titration at any dose | 1
Not completed — Less than 3 BTP episodes per week | 2
Period: Efficacy Phase
Arm/Group | Intranasal Fentanyl Spray (INFS)
Started | 15 (Participants titrated to 200 or 400 μg INFS in Titration Phase)
Completed | 13
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Death | 1
Period: Tolerability Phase
Arm/Group | Intranasal Fentanyl Spray (INFS)
Started | 31 (Participants entered directly from the Titration or Efficacy Phase)
Completed | 16
Not Completed | 15
Not completed — Death | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of INFS (including the initial test dose).
Arm/Group | Intranasal Fentanyl Spray (INFS)
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (9.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 46
Region of Enrollment [Number; unit: participants]
  Hungary | 33
  Norway | 10
  Russian Federation | 3
Site of Primary Tumour Reported in >5% Patients [Number; unit: participants]
  Breast | 14
  Lung respiratory system | 5
  Gastro-oesophageal | 1
  Colon/rectal | 3
  Pancreas | 6
  Female genital | 3
  Prostate | 3
  Urological | 7
  Unknown Primary Tumour | 2
  Liver | 1
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Pain Intensity Difference at 10 Minutes (PID10) After Treatment
Description: During the efficacy phase participants assessed their pain intensity at each breakthrough pain (BTP) episode at 0 and 10 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID10 is calculated as the difference in pain intensity from time 0 to 10 minutes. A positive value is a decrease (improvement) of the pain; a ≥ 2-point difference is considered as clinically important.
Time Frame: During the efficacy phase (II), at each episode of breakthrough pain, at 0 and 10 minutes after first dose of study drug.
Population: The Full Analysis Set consisted of all randomly assigned participants who entered the Efficacy Phase (II) of the trial and were treated for at least 1 BTP episode with double-blind INFS in the Efficacy Phase of the trial.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intranasal Fentanyl Spray (INFS): In the Efficacy phase participants received 400 μg INFS for 6 episodes of breakthrough pain.
- Placebo: In the Efficacy Phase Participants received placebo intranasal spray for 2 episodes of breakthrough pain.
Arm/Group | Intranasal Fentanyl Spray (INFS) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 2.5 [1.42 to 3.49] | 1.4 [0.23 to 2.48]
Statistical Analysis 1: Comparison: Intranasal Fentanyl Spray (INFS) vs Placebo; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; A mixed effects model with episode baseline PI as a covariate, treatment as a fixed effect and patient as a random effect; LS Mean Difference = 1.1, 95% CI 2-sided [0.41 to 1.179]

2. Secondary Outcome: Incidence of Improvement or Worsening in Nasal Mucosa Sign or Abnormality Score
Description: Medical examination of the nasal cavity by rhinoscopy was performed by an oto-rhino-laryngologist before the start of study treatment and at 12 weeks. Signs and any abnormalities were observed for each nostril using the following 4 points assessment scale: • 0 =not present; • 1 =present in a mild degree; • 2 =present in a moderate degree; • 3 =present in a severe degree. A difference in score of 1 or more from Baseline to the end of treatment represented a worsening, while a negative value indicated an improvement of the observed clinical sign. The oto-rhino-laryngologist also assessed whether worsening of a sign was related to study drug. Assessments for both left and right nostrils are presented together. The incidence is calculated as the number of assessments (n) in the improvement or worsening category divided by the number of assessments with a non-missing score for the Nasal Mucosa or Abnormality assessment. Only those signs or abnormalities with n>0 were included
Time Frame: Baseline and at 12 weeks
Population: Safety Analysis Set, which included all patients who received at least 1 dose of INFS (including the initial test dose) with non-missing assessments.
Measure: Number (95% Confidence Interval); unit: proportion of nostril assessments
Units Other Than Participants: Nostrils
Arm/Group | Intranasal Fentanyl Spray (INFS)
Number analyzed (Participants) | 46
Number analyzed (Nostrils) | 54
proportion of nostril assessments
  Change of color: Improvement | 0.06 [0.00 to 0.12]
  Change of color: Worsening | 0.09 [0.02 to 0.17]
  Change of color: Worsening related to study drug | 0.09 [0.02 to 0.17]
  Inflammation: Improvement | 0.04 [0.00 to 0.09]
  Inflammation: Worsening | 0.07 [0.00 to 0.14]
  Inflammation: Worsening related to study drug | 0.07 [0.00 to 0.14]
  Sore nose: Improvement | 0.04 [0.00 to 0.09]
  Sore nose: Worsening | 0.04 [0.00 to 0.09]
  Sore nose: Worsening related to study drug | 0.04 [0.00 to 0.09]
  Ulceration: Improvement | NA [NA to NA] — No participants achieved ulceration improvement.
  Ulceration: Worsening | 0.04 [0.00 to 0.09]
  Ulceration: Worsening related to study drug | 0.04 [0.00 to 0.09]
  Dry nose: Improvement | 0.09 [0.02 to 0.17]
  Dry nose: Worsening | 0.06 [0.00 to 0.12]
  Dry nose: Worsening related to study drug | NA [NA to NA] — No participants achieved worsening of dry nose related to study drug.
  Runny nose: Improvement | 0.04 [0.00 to 0.09]
  Runny nose: Worsening | 0.13 [0.04 to 0.22]
  Runny nose: Worsening related to study drug | 0.10 [0.02 to 0.18]
  Stuffed nose: Improvement | 0.06 [0.00 to 0.12]
  Stuffed nose: Worsening | 0.17 [0.07 to 0.27]
  Stuffed nose: Worsening related to study drug | 0.08 [0.00 to 0.15]
  Oedema: Improvement | 0.04 [0.00 to 0.09]
  Oedema: Worsening | 0.17 [0.07 to 0.27]
  Oedema: Worsening related to study drug | 0.08 [0.00 to 0.15]
  Epistaxis: Improvement | 0.02 [0.00 to 0.05]
  Epistaxis: Worsening | 0.02 [0.00 to 0.05]
  Epistaxis: Worsening related to study drug | 0.02 [0.00 to 0.05]

3. Secondary Outcome: Efficacy Phase: Pain Intensity Difference (PID) at 5, 30, and 60 Minutes After First Dose of Study Drug
Description: During the efficacy phase participants assessed their pain intensity at each breakthrough pain (BTP) episode at 0, 5, 30 and 60 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID is calculated as the difference in pain intensity from time 0 to each time point. A positive value is a decrease (improvement) of the pain; a ≥ 2-point difference is considered as clinically important.
Time Frame: During the efficacy phase (II) each episode of breakthrough pain, at 0, 5, 30 and 60 minutes after study drug.
Population: Efficacy Phase, Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intranasal Fentanyl Spray (INFS) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  PID at 5 minutes | 1.3 [0.72 to 1.89] | 0.8 [0.18 to 1.51]
  PID at 30 minutes | 3.0 [2.03 to 3.88] | 1.8 [0.79 to 2.88]
  PID at 60 minutes | 3.3 [2.34 to 4.17] | 2.2 [1.17 to 3.27]

4. Secondary Outcome: Efficacy Phase: Sum of Pain Intensity Differences (SPID0-60 and SPID0-30) Derived From PI Scores
Description: The SPID30 and SPID60 represent the average improvement in pain intensity over the 30 minute interval and 60 minute interval, respectively. SPIDt was calculated as the area under the curve (AUC) for Pain Intensity Difference over the time interval 0 to t minutes, respectively, divided by the length of the time interval (t minutes). A positive value is a decrease (improvement) of the pain.
  Pain intensity was assessed at 0, 5, 30 and 60 minutes after study drug using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID is calculated as the difference in pain intensity from time 0 to each time point.
Time Frame: During the efficacy phase (II) each episode of breakthrough pain, at 0, 5, 30 and 60 minutes after study drug
Population: Efficacy Phase, Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intranasal Fentanyl Spray (INFS) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale
  SPID30 | 0.6 [0.38 to 0.90] | 0.4 [0.09 to 0.67]
  SPID60 | 0.7 [0.46 to 1.04] | 0.5 [0.13 to 0.77]

5. Secondary Outcome: Efficacy Phase: Proportion of BTP Episodes With a Positive Response Defined as a ≥ 1, 2 or 3 Point Reduction in Pain Intensity
Description: Overall responder rate is defined as the proportion of breakthrough pain (BTP) episodes with a positive response to treatment. The following definitions of a positive response were analyzed: • greater than or equal to 1 point reduction in pain intensity (PI) from time 0, • greater than or equal to 2 point reduction in PI from time 0, and • greater than or equal to 3 point reduction in PI from time 0. Pain intensity was assessed using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain".
Time Frame: During the efficacy phase (II) each episode of breakthrough pain, at 0, 5, 30 and 60 minutes after study drug
Population: Efficacy Phase, Full Analysis Set
Measure: Number; unit: proportion of breakthrough pain episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Intranasal Fentanyl Spray (INFS) | Placebo
Number analyzed (Participants) | 15 | 15
Number analyzed (breakthrough pain episodes) | 88 | 29
proportion of breakthrough pain episodes
  ≥ 1 point reduction in PI at 5 minutes | 0.61 | 0.45
  ≥ 1 point reduction in PI at 10 minutes | 0.74 | 0.55
  ≥ 1 point reduction in PI at 30 minutes | 0.81 | 0.66
  ≥ 1 point reduction in PI at 60 minutes | 0.86 | 0.69
  ≥ 2 point reduction in PI at 5 minutes | 0.33 | 0.24
  ≥ 2 point reduction in PI at 10 minutes | 0.51 | 0.31
  ≥ 2 point reduction in PI at 30 minutes | 0.60 | 0.41
  ≥ 2 point reduction in PI at 60 minutes | 0.65 | 0.48
  ≥ 3 point reduction in PI at 5 minutes | 0.18 | 0.17
  ≥ 3 point reduction in PI at 10 minutes | 0.32 | 0.24
  ≥ 3 point reduction in PI at 30 minutes | 0.45 | 0.34
  ≥ 3 point reduction in PI at 60 minutes | 0.50 | 0.48

6. Secondary Outcome: Efficacy Phase: Proportion of BTP Episodes With a Positive Response Defined as a ≥ 33% or 50% Reduction in Pain Intensity
Description: Overall responder rate is defined as the proportion of breakthrough pain (BTP) episodes with a positive response to treatment. The following definitions of a positive response were analyzed: • Greater than 33% reduction in PI from time 0; • Greater than or equal to 50% reduction in PI from time 0. Pain intensity was assessed using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain".
Time Frame: During the efficacy phase (II) each episode of breakthrough pain, at 0, 5, 30 and 60 minutes after study drug
Population: Efficacy Phase, Full Analysis Set
Measure: Number; unit: proportion of breakthrough pain episodes
Units Other Than Participants: breakthrough pain episodes
Arm/Group | Intranasal Fentanyl Spray (INFS) | Placebo
Number analyzed (Participants) | 15 | 15
Number analyzed (breakthrough pain episodes) | 88 | 29
proportion of breakthrough pain episodes
  > 33% reduction in PI at 5 minutes | 0.23 | 0.17
  > 33% reduction in PI at 10 minutes | 0.44 | 0.24
  > 33% reduction in PI at 30 minutes | 0.55 | 0.34
  > 33% reduction in PI at 60 minutes | 0.58 | 0.48
  ≥ 50% reduction in PI at 5 minutes | 0.11 | 0.07
  ≥ 50% reduction in PI at 10 minutes | 0.31 | 0.21
  ≥ 50% reduction in PI at 30 minutes | 0.49 | 0.31
  ≥ 50% reduction in PI at 60 minutes | 0.52 | 0.34

7. Secondary Outcome: Efficacy Phase: General Impression (GI) Score at 60 Minutes After First Dose
Description: Participants assessed their general impression (GI) of treatment efficacy for treated BTP episodes at 60 minutes after first dose of study drug. The validated, categorical 5-point Verbal Rating Scale (VRS) was used for this assessment and scored as follows:
  * 0 =poor;
  * 1 =fair;
  * 2 =good;
  * 3 =very good;
  * 4 =excellent.
Time Frame: During the efficacy phase (II), at each episode of breakthrough pain, 60 minutes after first dose of study drug.
Population: Efficacy Phase, Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intranasal Fentanyl Spray (INFS) | Placebo
Number analyzed (Participants) | 15 | 15
units on a scale | 1.9 [1.41 to 2.47] | 1.1 [0.52 to 1.71]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The severity (intensity of each AE was assessed as mild (transient symptoms, no interference with daily activities), moderate (marked symptoms, moderate interference with daily activities), or severe (considerable interference with daily activities) by the investigator. Serious adverse events are defined as any untoward medical occurrence that at any dose results in death or is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect. The investigator assessed each AE as either related or not related to study treatment.
Time Frame: 12 weeks
Population: Safety analysis set
Measure: Number; unit: participants
Groups:
- Titration Phase: All participants were step-wise titrated to an effective dose of 50, 100, 200 or 400 μg INFS in the Titration Phase.
- Efficacy Phase: Participants titrated to 200 or 400 μg INFS in the Titration Phase were randomized to an 8-spray sequence in the Efficacy Phase (II); 6 BTP episodes were treated with 400 μg INFS and 2 BTP episodes with placebo in a random sequence.
- Tolerability Phase: Participants entered the Tolerability Phase (III) either directly from the Titration Phase (with an effective dose of 50 or 100 μg) or from the Efficacy Phase (400 μg) and continued with this specific dose, unless adjustment was needed, for a total treatment time of 12 weeks.
Arm/Group | Titration Phase | Efficacy Phase | Tolerability Phase
Number analyzed (Participants) | 45 | 15 | 31
participants
  Any AE | 23 | 6 | 22
  Any AE reported as related to treatment | 14 | 4 | 6
  Non-serious adverse events | 22 | 5 | 17
  Serious adverse events | 2 | 2 | 8
  Deaths | 2 | 1 | 5
  Severe adverse events | 2 | 2 | 7
  AEs leading to withdrawal | 2 | 2 | 3
  AEs possibly associated with nasal intolerability | 2 | 0 | 6
  AEs with an onset within 30 minutes of first dose | 11 | 3 | 5

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Titration Phase: Participants were step-wise titrated to an effective dose of 50, 100, 200 or 400 μg INFS in the Titration Phase (I).
Arm/Group | Titration Phase | Efficacy Phase | Tolerability Phase
Serious Adverse Events (participants affected / at risk) | 2/45 | 2/15 | 8/31
Other Adverse Events (participants affected / at risk) | 22/45 | 5/15 | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Titration Phase (N=45) | Efficacy Phase (N=15) | Tolerability Phase (N=31)
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1 | 0
Device occlusion (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Titration Phase (N=45) | Efficacy Phase (N=15) | Tolerability Phase (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 10 | 1 | 8
Vomiting (Gastrointestinal disorders) | 3 | 1 | 4
Asthenia (General disorders) | 1 | 0 | 1
Discomfort (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 1
General physical health deterioration (General disorders) | 2 | 0 | 1
Irritability (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 8 | 2 | 4
Headache (Nervous system disorders) | 1 | 0 | 3
Horner's syndrome (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Sedation (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Emotional distress (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.